CLINICAL TRIAL: NCT06461169
Title: The Effect of Stress Ball on Pain, Anxiety and Physiological Parameters in COPD Patients Receiving Noninvasive Mechanical Ventilation Support
Brief Title: The Effect of Stress Ball on COPD Patients Receiving Noninvasive Mechanical Ventilation Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Huseyin Seker, nurse, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KafkasUniversity
Record Dates: First submitted 2024-05-09; First posted 2024-06-14 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: COPD; COPD Exacerbation
Keywords: anxiety; pain; CPAP; vital signs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Block randomisation will be used to ensure that the number of patients in each group is balanced. Patients will be divided into two groups, each group consisting of at least 30 people, by a statistician who is not involved in the study, using a table of random numbers.
Who Masked: Outcomes Assessor
Masking Description: In the study, blinding will be performed only in the assignment-randomisation to groups and statistical analysis of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional (Experimental): group applying the stress ball during the CPAP procedure
  Interventions: Other: stress ball
- control (No Intervention): The group in which no intervention was carried out and the routine care was provided by the nurses during the CPAP procedure

INTERVENTIONS:
Other: stress ball — Patients squeeze the stress ball
  Arms: interventional

SUMMARY:
The aim of this randomised controlled trial was to investigate the effect of a stress ball on pain, anxiety and physiological parameters in Chronic Obstructive Pulmonary Disease (COPD) patients on non-invasive mechanical ventilation (NIMV).

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure (CPAP) therapy used in NIMV reduces the need for IMV in COPD patients and shortens hospital stays. Negative states resulting from the difficulty of treatment lead to increased pain and anxiety in patients and negative results in vital signs. There is a need for non-invasive, low-cost and easy-to-use methods that can be used by nurses to address these problems in patients. This study will investigate the effect of a stress ball on changes in pain, anxiety and vital signs in patients diagnosed with COPD and receiving CPAP treatment during treatment. The stress ball will be applied to the patients during two consecutive CPAP treatments and pain, anxiety scores and vital signs will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD
* Receiving CPAP therapy
* Those who voluntarily agreed to participate in the study
* Turkish speaking, understanding,
* No cognitive and cognitive problems
* glasgow coma scale score of 13 and above
* Those who have not participated in stress ball etc. application before

Exclusion Criteria:

* Refused to participate in the research
* People with visual and hearing impairment
* unable to speak and understand Turkish
* Cognitive and cognitive problems
* glasgow coma scale<13
* Infection, wound, burn, plaster, traction etc. in the hand and arm area
* During the research, those who wanted to leave voluntarily
* General condition deteriorated during NIMV treatment

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
face anxiety scale | Change in anxiety score at the beginning of the intervention and 1 hour later
  Developed in 2003, the Facial Anxiety Scale is a measurement tool in which patients self-report their anxiety levels and is 11 × 42 cm in size. It consists of five face shapes, the leftmost facial expression indicates the absence of anxiety, while the level of anxiety increases towards the right (scored between 0-5). According to the Facial Anxiety Scale, a score of 3 and above by the patients indicates that the level of anxiety is at medium and high levels.
Visual Analogue Scale (Pain) Visual analog scale (VAS) | Change in pain score at the beginning of the intervention and 1 hour later
  Visual analog scale is used to convert parameters that cannot be measured numerically into a numerical value. For pain, '0: I have no pain and 10: I have unbearable/severe pain' is written on one end of a 100 mm line and the patient marks his/her current condition on this line.

SECONDARY OUTCOMES:
systolic blood pressure (mm/Hg) | at the beginning of the intervention and at the 15th, 30th, 45th and 60th minutes of the intervention
  the effect of the intervention on systolic blood pressure is examined
diastolic blood pressure (mm/Hg) | at the beginning of the intervention and at the 15th, 30th, 45th and 60th minutes of the intervention
  the effect of the intervention on diastolic blood pressure is examined
SpO2-peripheral oxygen saturation (%) | at the beginning of the intervention and at the 15th, 30th, 45th and 60th minutes of the intervention
  the effect of the intervention on peripheral oxygen saturation is examined
respiratory rate (minute value) | at the beginning of the intervention and at the 15th, 30th, 45th and 60th minutes of the intervention
  the effect of the intervention on respiratory rate is examined
heart rate (minute value) | at the beginning of the intervention and at the 15th, 30th, 45th and 60th minutes of the intervention
  the effect of the intervention on heart rate is examined

CONTACTS AND LOCATIONS:
Locations (1):
- Kafkas University, Kars, Merkez, Turkey (Türkiye)